CLINICAL TRIAL: NCT04849065
Title: Clinical Trial in Phase II of Intramuscular Infusion of Autologous Bone Marrow Stem Cells in Patients With Amyotrophic Lateral Sclerosis.
Brief Title: Clinical Trial on the Use of Cell Therapy in the Treatment of Patients With Amyotrophic Lateral Sclerosis
Acronym: TCIM-ELAII
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Fundacion para la Formacion e Investigacion Sanitarias de la Region de Murcia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IMB-TCIM/ELAII-2019-01
Record Dates: First submitted 2021-04-15; First posted 2021-04-19 (Actual); Last update posted 2021-04-19 (Actual); Status verified 2021-04

CONDITIONS: ALS (Amyotrophic Lateral Sclerosis)
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis | interventions — Sodium Chloride

STUDY DESIGN:
Intervention Model Description: Phase II, prospective, multicenter, randomized, parallel, double-blind, placebo-controlled clinical trial
Who Masked: Participant, Investigator
Masking Description: double-blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MNC (Mononuclear cells) (Experimental): MNC (Mononuclear cells) (patients in which stem cells will be injected into the two muscles on one side and placebo -vehicle- in the two contralateral muscles).
  This group would consist of 74 patients.
  Interventions: Drug: MNC (Mononuclear cells); Drug: Placebo / Saline
- Saline (Placebo Comparator): (patients in which placebo -vehicle- will be injected into both muscles on both sides). This group would consist of 26 patients.
  Interventions: Drug: Placebo / Saline

INTERVENTIONS:
Drug: MNC (Mononuclear cells) — * Intramuscular infusion of autologous BM CMN into the TA muscle of one of the lower limbs (experimental side)
  * Intramuscular infusion of saline solution (placebo) in the TA muscle of the contralateral lower limb (control side)
  Arms: MNC (Mononuclear cells)
Drug: Placebo / Saline — - Intramuscular infusion of saline solution (placebo) in the TA muscle of the contralateral lower limb (control side)

SUMMARY:
Our working hypothesis is that the injection of autologous bone marrow mononuclear cells (BMNC) has a positive effect on the natural loss of motor units and on the increase in the size of the motor unit that occurs in patients with ALS during the evolution of the disease

DETAILED DESCRIPTION:
Our working hypothesis is that the injection of autologous bone marrow mononuclear cells (BMNC) has a positive effect on the natural loss of motor units and on the increase in the size of the motor unit that occurs in patients with ALS during the evolution of the disease.

This hypothesis is based on experimental work done in animal models of ALS and the results of our previous phase I clinical trial. In this clinical trial (TCIM / ALS, ClinicalTrials.gov Identifier: NCT02286011) we studied with electrophysiological techniques (in a small number of patients with ALS) the effects of intramuscular injection of a single dose of BMSC in the tibialis anterioris (TA) muscle. . The results indicate that this is a safe procedure and show the presence of a positive and apparently transitory effect on the size and number of motor units of the TA muscle.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of ALS defined or probable according to the criteria established by the World Federation of Neurology
* Age between 18 and 70 years.
* Patient who offers sufficient guarantees of adherence to the protocol.
* Neurophysiological data confirming lower motor neuron involvement at the lumbar and cervical level.
* Assessment of the motor deficit in the dorsal flexion of both feet (between 3 and 5 points on the MRC scale).

Exclusion Criteria:

* Mellitus diabetes.
* Other diseases that may be associated with polyneuropathies.
* Previous history of cerebral stroke.
* Previous pathology of the peripheral nervous system that affected one or both lower or upper limbs, with or without clinically evident neurological sequelae.
* Pregnant or actively breastfeeding patients
* Patients physiologically capable of becoming pregnant, unless they are using a reliable contraceptive method (Annex III)
* Patients with cardiac, renal, hepatic, systemic, immune disease that may influence the survival of the patient during the test.
* Positive serology for hepatitis B, hepatitis C or HIV.
* Clinical and anesthesiological criteria that contraindicate either sedation or the extraction of BM itself (Alteration of the coagulation system or anticoagulated patient with inability to withdraw anticoagulation, hemodynamic instability, skin alteration in the puncture site, etc.)
* Inclusion in other clinical trials in the last 6 months.
* Inability to understand informed consent.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2021-05-01 (Estimated); Primary Completion 2023-05-01 (Estimated); Study Completion 2023-09-01 (Estimated)

PRIMARY OUTCOMES:
Rate of serious and non-serious adverse events related to the use of bone marrow mononuclear cells in patients with Amyotrophic Lateral Sclerosis | 48 months from baseline
D50 index obtained from stimulus intensity curves | 48 months from baseline
  This parameter quantifies the number and size of the functional motor units of a given muscle.

SECONDARY OUTCOMES:
Motor unit number index" (MUNIX) | 48 months from baseline
  The unit amplitude (or area) of the individual motor units are calculated from the amplitude variations (or area) of the muscle action potential obtained in response to stimuli from a fixed intensity
Motor unit size index" (MUSIX) | 48 months from baseline
  The unit amplitude (or area) of the individual motor units are calculated from the amplitude variations (or area) of the muscle action potential obtained in response to stimuli from a fixed intensity
Fiber density (FD) | 48 months from baseline
  Quantifies the average number of muscle fibers per motor unit. It is obtained from single fiber recordings made with electrodes. The average number of motor unit potentials is calculated in 20 different positions in the muscle.
PAMC amplitude: mV | 48 months from baseline
  Compound muscle action potential (CMAP)
PAMC area: mV / ms | 48 months from baseline
  Compound muscle action potential (CMAP)
Maximum force developed in an isometric contraction of the muscles | 48 months from baseline
  The measurement will be made with a dynamometer during dorsiflexion of the foot (from certain angles) and during abduction of the index finger of the hand, respectively.
Fuerza muscular (MRC Medical Research Council) score | 48 months from baseline
  Muscle strength data will be collected according to the Medical Research Council scale. Muscle strength is graded on a scale of 0 to 5, with 5 being normal muscle strength and 0 being the absence of muscle contraction.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Clinico Universitario Virgen de la Arrixaca, Murcia, Spain

IPD SHARING:
Plan to Share IPD: No